CLINICAL TRIAL: NCT02299973
Title: Fecal Microbiota Transplantation in Irritable Bowel Syndrome With Bloating: a Double Blind, Placebo Controlled Randomised Clinical Trial
Brief Title: Fecal Microbiota Transplantation in Irritable Bowel Syndrome With Bloating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Gastro-enterologie, Gastro-enterologie, University Hospital, Ghent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGent_Gastro_001
Record Dates: First submitted 2014-11-11; First posted 2014-11-24 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; fecal microbiota transplantation; bloating
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (FMT with own stool) (Placebo Comparator): Fecal microbiota transplantation with patient's own stool
  Interventions: Procedure: FMT with own stool
- Treatment group (FMT with donor stool) (Experimental): Fecal microbiota transplantation with healthy donor stool
  Interventions: Procedure: FMT with donor stool

INTERVENTIONS:
Procedure: FMT with donor stool — fecal microbiota transplantation by means of colonoscopy with deliverance of the transplant in the right colon and terminal ileum. Transplants will be collected prior to the start of the study from a healthy pool of donors and will be frozen at -80 degrees celsius after thorough screening for infectious diseases. At the time of transplantation samples will be frozen and administrated to the patients in the treatment group
  Other Names: Fecal microbiota transplantation with healthy donor stool
  Arms: Treatment group (FMT with donor stool)
Procedure: FMT with own stool — fecal microbiota transplantation by means of colonoscopy with deliverance of the transplant in the right colon and terminal ileum. Transplants will be collected prior to the start of the study from the patients and will be frozen at -80 degrees celsius after thorough screening for infectious diseases. At the time of transplantation samples will be frozen and administrated to the patients in the control group
  Other Names: Fecal microbiota transplantation with own stool
  Arms: Placebo group (FMT with own stool)

SUMMARY:
Intestinal microbiota dysbiosis is thought to play an important role in the complex pathophysiology of irritable bowel syndrome (IBS), especially in diarrhoea-predominant IBS and possibly in IBS with severe bloating. Fecal microbiota transplantation or FMT has been shown to be an effective means of correcting this imbalance in the gut microbiota, especially in patients with recurrent Clostridium difficile infections where it has become a preferred treatment strategy.

In a preliminary pilot study in 12 patients we found that FMT was a safe and accepted therapy in IBS patients. In 75% of patients an amelioration of IBS symptoms in general and abdominal bloating was seen three months after transplantation.

In this study the effects of FMT on patients with IBS without constipation and bloating will be investigated in a double blind, placebo controlled RCT.

DETAILED DESCRIPTION:
Intestinal microbiota dysbiosis is thought to play an important role in the complex pathophysiology of irritable bowel syndrome (IBS), especially in diarrhoea-predominant IBS and possibly in IBS with severe bloating. Fecal microbiota transplantation or FMT has been shown to be an effective means of correcting this imbalance in the gut microbiota, especially in patients with recurrent Clostridium difficile infections where it has become a preferred treatment strategy.

In a preliminary pilot study in 12 patients we found that FMT was a safe and accepted therapy in IBS patients. In 75% of patients an amelioration of IBS symptoms in general and abdominal bloating was seen three months after transplantation.

In this study the effects of FMT on patients with IBS without constipation and bloating will be investigated in a double blind, placebo controlled RCT. Donors for this study will be recruited from a healthy donor pool who will donate stool after clearance of a strict inclusion protocol which will assess the presence of any infectious diseases. Stool will be frozen following the protocol described in Hamilton et al 2012. Patients will deliver a stool portion that will be frozen as well.

At time of FMT, patients will be randomised in a double blinded fashion to the treatment arm (healthy donor stool) or placebo arm (own stool). Transplantation will be preformed by means of a colonoscopy with deliverance in the right colon and ileum.

Following FMT patients will be followed clinically with questionnaires and regular visits to the clinic. Stool samples will be collected on a regular basis for microbiome analysis.

At the end of the study, patients from the placebo-group will be given the opportunity to be transplanted with healthy donor stool if necessary. Follow-up will continu for a total duration of one year.

ELIGIBILITY:
1. Inclusion Criteria for patients:

   * signed informed consent
   * Irritable bowel syndrome with predominant diarrhoea as defined by the ROME III criteria and with symptoms of abdominal bloating
   * IBS symptom score > 3 on at least 2 subscores (abdominal discomfort, abdominal bloating, abdominal pain, urgency, stool frequency, stool consistency)
2. Exclusion Criteria for patients:

   * predominant constipation as defined by Rome III criteria
   * pregnancy or inadequate anti conception for the duration of the trial
   * celiac disease
   * any contra-indications for colonoscopy
   * structural abnormalities of the colon (e.g. ileocecal resection, gastric bypass)
   * severe gastro-intestinal comorbidities (e.g. IBD, coloncarcinoma)
   * non gastro-intestinal malignancy
   * severe psychiatric comorbidity which had important effects on the quality of life
   * antimicrobial treatment 4 weeks prior to screening visit
   * treatment with probiotics 2 weeks prior to screening visit
   * recent diagnosis of lactose intolerance (< 3 months before screening visit)
   * any severe comorbidity that might interfere with the study course as determined by the treating physician
3. Inclusion criteria for donors

   * age 18 - 75 years
   * signed informed consent
   * normal screening protocol which includes screening for infectious diseases (eg. blood HIV, Syphilis, Hepatitis B or C; stool: enteropathogens, clostridium, ESBL, CPE)
4. Exclusion criteria for donors

   * presence of gastrointestinal symptoms
   * gastro-intestinal or other important comorbidity
   * obesity or metabolic syndrome
   * history of malignancy both gastrointestinal or systemic
   * presence of known colon polyps
   * recent placing of piercings/tattoos
   * sexual risk behaviour
   * antimicrobial therapy 3 months prior to donation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Reduction of overall IBS symptoms (Key question 1) | 3 months after FMT
  On a weekly basis patients will assess their overall IBS symptoms by answering a key question (Are your overall symptoms improved as compared to before the treatment?)
Reduction of abdominal bloating (Key question 2) | 3 months after FMT
  On a weekly basis patients will assess their sensation of abdominal bloating by answering a key question (Is your overall sensation of bloating improved by FMT as compared to before treatment?)

SECONDARY OUTCOMES:
Changes in fecal microbiome composition (Illumina sequencing) | 3 months after FMT
  Before and after FMT stool samples will be collected on a regular basis to assess the changes in microbiome changes (Illumina sequencing).
Changes in IBS symptom scores at three months after FMT | 3 months after FMT
  IBS symptoms will be assessed by use of a daily symptom diary which will measure abdominal discomfort, pain, bloating, flatulence, stool frequency, stool consistency and urgency
Changes in IBS symptom scores at six months post FMT | 6 months
  Key questions and symptom diary scores will be repeated 6 months after FMT to assess the duration of effects
Changes in IBS symtom scores at 9 months post FMT | 9 months
  Key questions and symptom diary scores will be repeated 9 months after FMT to assess the duration of effects
Changes in IBS symptom scores at 1 year post FMT | 1 year
  Key questions and symptom diary scores will be repeated 1 year after FMT to assess the duration of effects
Composition of mucosal-adherent microbiota (Illumina sequencing) | 3 months
  Composition of mucosal-adherent microbiota will be assessed by Illumina sequencing. Biopsies will be taken at time of FMT and snap frozen for further analysis.
Changes of IBS symptom scores in patients who undergo an off-trial FMT | 3 months
  After unblinding patients who were included in the placebo group, will be offered the possibility of FMT. Effects in these patients will be followed by IBS symptoms scores and answers to key questions at 3 months post FMT

CONTACTS AND LOCATIONS:
Overall Officials: Danny De Looze, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Background] Dupont HL. Review article: evidence for the role of gut microbiota in irritable bowel syndrome and its potential influence on therapeutic targets. Aliment Pharmacol Ther. 2014 May;39(10):1033-42. doi: 10.1111/apt.12728. Epub 2014 Mar 25. PMID 24665829
- [Background] Kassinen A, Krogius-Kurikka L, Makivuokko H, Rinttila T, Paulin L, Corander J, Malinen E, Apajalahti J, Palva A. The fecal microbiota of irritable bowel syndrome patients differs significantly from that of healthy subjects. Gastroenterology. 2007 Jul;133(1):24-33. doi: 10.1053/j.gastro.2007.04.005. Epub 2007 Apr 14. PMID 17631127
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Borody TJ, Paramsothy S, Agrawal G. Fecal microbiota transplantation: indications, methods, evidence, and future directions. Curr Gastroenterol Rep. 2013 Aug;15(8):337. doi: 10.1007/s11894-013-0337-1. PMID 23852569
- [Derived] Holvoet T, Joossens M, Vazquez-Castellanos JF, Christiaens E, Heyerick L, Boelens J, Verhasselt B, van Vlierberghe H, De Vos M, Raes J, De Looze D. Fecal Microbiota Transplantation Reduces Symptoms in Some Patients With Irritable Bowel Syndrome With Predominant Abdominal Bloating: Short- and Long-term Results From a Placebo-Controlled Randomized Trial. Gastroenterology. 2021 Jan;160(1):145-157.e8. doi: 10.1053/j.gastro.2020.07.013. Epub 2020 Jul 15. PMID 32681922